CLINICAL TRIAL: NCT02552888
Title: Nitrite, Isoquercetin and Endothelial Dysfunction (NICE) Trial
Acronym: NICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TulaneU; 1U54GM104940 (NIH)
Record Dates: First submitted 2015-09-10; First posted 2015-09-17 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Chronic Kidney Disease
Keywords: Endothelial Dysfunction; Inflammation; Oxidative Stress; eGFR; Urine Albumin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — isoquercitrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): Immediate release sodium nitrite 40 mg by mouth twice per day and Isoquercetin 225 mg by mouth once per day.
  Interventions: Drug: Immediate release sodium nitrite; Dietary Supplement: Isoquercetin
- Placebos (Placebo Comparator): identical placebos.
  Interventions: Other: placebos

INTERVENTIONS:
Drug: Immediate release sodium nitrite — Immediate release sodium nitrite 40 mg by mouth twice per day
  Other Names: TV1001
  Arms: treatment
Dietary Supplement: Isoquercetin — Isoquercetin 225 mg by mouth once per day
  Other Names: 3-O-glucoside
  Arms: treatment
Other: placebos — placebos
  Arms: Placebos

SUMMARY:
The proposed randomized controlled trial will test the safety and efficacy of combination therapy with sodium nitrite and isoquercetin on endothelial function and inflammation among patients with chronic kidney disease.

DETAILED DESCRIPTION:
The proposed randomized controlled trial will test the safety and efficacy of combination therapy with sodium nitrite and isoquercetin on endothelial function and inflammation among patients with chronic kidney disease. Investigators will recruit 70 albuminuric CKD patients and randomly assign participants to combination therapy with sodium nitrite and isoquercetin or placebo for three months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 21-74 years old with any race/ethnicity background
* CKD as defined by an eGFR <60 ml/min/1.73 m2 or urinary albumin to creatinine ratio ≥ 30 mg/g or protein to creatinine ratio ≥150 mg/g.
* Systolic BP≥120 and <180 mmHg and/or diastolic BP≥70 and <110 mmHg

Exclusion Criteria:

* Allergic to organic nitrite, isoquercetin, niacin, or vitamin C
* Institutionalized (e.g., prisoner, nursing home or skilled nursing facility resident)
* Unable or unwilling to give consent
* Known HIV infection and/or AIDS
* Pregnant or lactating women
* Currently on dialysis
* Previous or current organ or bone marrow transplant
* Receiving immunosuppressive treatment or other immunotherapy
* Receiving chemotherapy or alkylating agents for systemic cancer
* Recent acute myocardial infarction, cerebrovascular accidence or transient ischemic attack, or hospitalization in 3 months
* Acute kidney injury within the previous 3 months
* Currently taking a phosphodiesterase-5 enzyme inhibitor, such as Viagra
* History of chronic headaches
* Chronically receiving fluoroguinolones, cyclosporin (neural, sandimmune), nitrate drug, NSAIDS ( except aspirin ≤ 81 mg daily), allopurinol or uloric, meperidine and related central nervous system (CNS) depressants, oral glucocorticoids, and not willing or able to stop during study period.
* Active infection (i.e. systemic or osteomyelitis)
* Class III or IV heart failure
* History of hemolytic anemia including sickle cell disease
* Hemoglobin <10
* History of chronic obstructive pulmonary disease (COPD)
* Have a positive screen for glucose-6-phosphate dehydrogenase (G6PD) deficiency at screening
* Involvement in other clinical trials
* Current alcohol or other substance abuse
* Current smokers
* Unwillingness to stop flavonoid supplementation
* Unwillingness to stop nitrate and/or nitrite supplementation

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity.
Enrollment: 70 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane School of Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
deidentified data sets may be available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: no end date.
Access Criteria: The de-identified patient level data will be provided directly to the researcher in a secure manner, and the researcher is responsible for protecting the confidentiality and integrity of the data while the research is conducted.

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Chen J, Hamm LL, Bundy JD, Kumbala DR, Bodana S, Chandra S, Chen CS, Starcke CC, Guo Y, Schaefer CM, Lustigova E, Mahone E, Vadalia AM, Livingston T, Obst K, Hernandez J, Bokhari SR, Kleinpeter M, Alper AB, Lukitsch I, He H, Nieman DC, He J. Combination Treatment with Sodium Nitrite and Isoquercetin on Endothelial Dysfunction among Patients with CKD: A Randomized Phase 2 Pilot Trial. Clin J Am Soc Nephrol. 2020 Nov 6;15(11):1566-1575. doi: 10.2215/CJN.02020220. Epub 2020 Oct 6. PMID 33023894

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Placebos
Started | 35 (35 participants were enrolled.) | 35 (35 participants were enrolled.)
Completed | 34 (34 participants completed the study.) | 34 (34 participants completed the study)
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebos | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.4) | 62.2 (10.2) | 61.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 22 | 22 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 15 | 32
  White | 16 | 20 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Baseline Characteristics of Study Participants by Treatment Allocation
  participants
    United States | 35 | 35 | 70
Baseline Metabolic Panel of Study Participants by Treatment Allocation [Mean (Standard Deviation); unit: mg/dL]
  Fasting plasma glucose, mean, mg/dL | 119 (44) | 124 (70) | 121.5 (57)
  Total cholesterol, mean, mg/dL | 178 (43) | 171 (50) | 174.5 (46.5)
  HDL-cholesterol, mean, mg/dL | 48 (13) | 47 (14) | 47.5 (13.5)
  LDL-cholesterol, mean, mg/dL | 107 (34) | 100 (37) | 103.5 (35.5)
Baseline Blood Pressure of Study Participants by Treatment Allocation [Mean (Standard Deviation); unit: mmHg]
  Systolic blood pressure, mean, mmHg | 129 (15) | 129 (15) | 129 (15)
  Diastolic blood pressure, mean, mmHg | 73 (7) | 75 (11) | 74 (9)
Baseline Body Mass Index of Study Participants by Treatment Allocation [Mean (Standard Deviation); unit: kg/m^2] | 30.9 (5.6) | 32.5 (5.7) | 31.7 (5.65)
Baseline Estimated Glomerular Filtration Rate of Study Participants by Treatment Allocation [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 51 (22) | 45 (16) | 48 (19)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change in Endothelium-dependent Flow-mediated Vasodilation (FMD) Over 12 Weeks
Description: FMD was measured using high resolution ultrasound on the brachial artery. FMD was calculated as the maximal percentage change in vessel size during hyperemia . The mean changes between baseline, 6 weeks and 12 weeks in FMD with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Treatment | Placebos
Number analyzed (Participants) | 35 | 35
Percentage change | 1.1 [-0.1 to 2.3] | 0.3 [-0.9 to 1.5]

2. Secondary Outcome: Mean Change in Endothelial Function Biomarkers VCAM-1, ICAM-1, E-selectin and vWF Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of Vascular Adhesion Molecule-1(VCAM-1), Intercellular Adhesion Molecule-1 (ICAM-1), E-selectin, and von Willebrand Factor (vWF). The mean changes between baseline, 6 weeks and 12 weeks in VCAM-1, ICAM-1, E-selectin and vWF with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Treatment: Immediate release sodium nitrite 40 mg by mouth twice per day and Isoquercetin 225 mg once daily
- Placebo: identical placebos
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
ng/mL
  ICAM, ng/mL | -16.1 [-41.5 to 9.3] | -4.0 [-29.0 to 21]
  VCAM-1, ng/mL | -22.2 [-49.3 to 5.0] | -10.8 [-37.5 to 15.9]
  E-Selecint, ng/mL | -0.32 [-3.14 to 2.50] | 1.06 [-1.73 to 3.84]
  vWF, ng/mL | -683 [-3784 to 2419] | 2744 [-328 to 5815]

3. Secondary Outcome: Mean Change in Endothelial Function Biomarker Asymmetrical DiMethylArginine (ADMA) Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of Asymmetrical DiMethylArginine (ADMA). The mean changes between baseline, 6 weeks and 12 weeks in ADMA with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: umol/mL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
umol/mL | 0.03 [-0.02 to 0.08] | 0.02 [-0.03 to 0.07]

4. Secondary Outcome: Mean Change in Endothelial Function Biomarker Endostatin Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of endostatin. The mean changes between baseline, 6 weeks and 12 weeks in endostatin with 95% CI were calculated using linear mixed effects model, and the log transformed endostatin was calculated.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: log (ng/mL)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
log (ng/mL) | -0.02 [-0.08 to 0.05] | -0.01 [-0.08 to 0.05]

5. Secondary Outcome: Mean Change in Endothelial Function Biomarker Urine Epidermal Growth Factor (UEGF) Over 12 Weeks
Description: A urine sample was taken for each participant to measure the levels of Urine Epidermal Growth Factor (UEGF). The mean changes between baseline, 6 weeks and 12 weeks in UEGF with 95% CI were calculated using linear mixed effects model, and the log transformed Urine EGF/creatinine ratio was calculated.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: log (pg/g)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
log (pg/g) | -0.01 [-0.39 to 0.37] | 0.23 [-0.14 to 0.61]

6. Secondary Outcome: Mean Change in Inflammatory Biomarker C-Reactive Protein (CRP) Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of C-Reactive Protein (CRP). The mean changes between baseline, 6 weeks and 12 weeks in CRP with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: mg/mL
Groups:
- Treatment: Immediate release sodium nitrite 40 mg by mouth twice per day and Isoquercetin 225 mg by mouth once daily
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
mg/mL | 0.05 [-0.31 to 0.42] | -0.02 [-0.38 to 0.33]

7. Secondary Outcome: Mean Change in Inflammatory Biomarkers Tumor Necrosis Factor-α (TNF-a), Interleukin-17 (IL-17), Interleukin-1β (IL-1beta), and Monocyte Chemoattractant Protein-1 (MCP-1) Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of Tumor Necrosis Factor-α (TNF-a), interleukin-17 (IL-17), interleukin-1β (IL-1beta), and Monocyte Chemoattractant Protein-1 (MCP-1). The mean changes between baseline, 6 weeks and 12 weeks in TNF-a, IL-17, IL-1beta, MCP-1 with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
pg/mL
  TNF-a, pg/mL | -0.04 [-0.20 to 0.12] | -0.04 [-0.20 to 0.12]
  IL-17, pg/mL | -0.72 [-1.80 to 0.36] | 0.01 [-1.05 to 1.08]
  IL-1 beta, pg/mL | -17.1 [-77.5 to 43.4] | -30.5 [-90.0 to 29.0]
  MCP-1, pg/mL | -6.0 [-25.0 to 13.0] | 0.6 [-18.0 to 19.3]

8. Secondary Outcome: Mean Change in Inflammatory Biomarker Interleukin-6 (IL-6) Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of interleukin-6 (IL-6). The mean changes between baseline, 6 weeks and 12 weeks in interleukin-6 (IL-6) with 95% CI were calculated using linear mixed effects model, and the log transformed IL-6 was calculated.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: log (pg/mL)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
log (pg/mL) | 0.07 [-0.06 to 0.20] | -0.17 [-0.30 to -0.04]

9. Secondary Outcome: Mean Change in Oxidative Stress Biomarker Low-density Lipoprotein (LDL) Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of low-density lipoprotein (LDL). The mean changes between baseline, 6 weeks and 12 weeks in LDL with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
ng/mL | -1.7 [-3.9 to 0.5] | -0.3 [-2.4 to 1.9]

10. Secondary Outcome: Mean Change in Oxidative Stress Biomarker Nitrotyrosine Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of nitrotyrosine. The mean changes between baseline, 6 weeks and 12 weeks in nitrotyrosine with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
pg/mL | -10.9 [-96.9 to 75.2] | 62.2 [-22.6 to 147.0]

11. Other Pre Specified Outcome: Mean Percentage Change in Methemoglobin Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of methemoglobin. The mean percentage change between baseline, 6 weeks and 12 weeks in methemoglobin with 95% CI was calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
Percentage change | -0.06 [-0.11 to -0.01] | -0.05 [-0.11 to -0.01]

12. Other Pre Specified Outcome: Mean Change in Isoquercetin Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of isoquercetin. The mean changes between baseline, 6 weeks and 12 weeks in isoquercetin with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: ug/L
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
ug/L | 166 [102 to 230] | 11.7 [-51.1 to 74.5]

13. Other Pre Specified Outcome: Mean Change in Plasma Nitrite Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of plasma nitrite. The mean changes between baseline, 6 weeks and 12 weeks in plasma nitrite with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: micromol/L
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
micromol/L | -0.07 [-0.20 to 0.05] | -0.11 [-0.23 to 0.01]

14. Other Pre Specified Outcome: Mean Change in Estimated-Glomerular Filtration Rate (eGFR) Over 12 Weeks
Description: Estimated-Glomerular Filtration Rate (eGFR) was calculated using the Chronic Kidney Disease Epidemiology Collaboration equation. The equation is GFR = 141 * min(Scr/κ,1)α * max(Scr/κ, 1)-1.209 * 0.993Age * 1.018 [if female] * 1.159 [if black]. Scr is serum creatinine (mg/dL), κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1. The mean changes between baseline, 6 weeks and 12 weeks in eGFR with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
mL/min/1.73 m^2 | 0.1 [-2.3 to 2.5] | 0.2 [-2.2 to 2.6]

15. Other Pre Specified Outcome: Mean Change in Lipid Profile Biomarkers Total Cholesterol, Low Density Lipoprotein (LDL)-Cholesterol and High Density Lipoprotein (HDL)-Cholesterol Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of total cholesterol, Low Density Lipoprotein (LDL)-cholesterol and High Density Lipoprotein (HDL)-cholesterol. The mean changes between baseline and 12 weeks in total cholesterol, Low Density Lipoprotein (LDL)-cholesterol and High Density Lipoprotein (HDL)-cholesterol with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline,12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
mg/dL
  Total Cholesterol, mg/dL | -1.6 [-10.5 to 7.2] | 3.9 [-4.9 to 12.8]
  LDL-cholesterol, mg/dL | -1.9 [-7.4 to 3.7] | 0.9 [-7.4 to 3.7]
  HDL-cholesterol, mg/dL | 0.9 [-1.7 to 3.4] | 2.2 [-0.4 to 4.7]

16. Other Pre Specified Outcome: Mean Change in Lipid Profile Biomarker Triglycerides Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of triglycerides. The mean changes between baseline and 12 weeks in triglycerides with 95% CI were calculated using linear mixed effects model, and the log transformed triglyceride was calculated.
Time Frame: Baseline,12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: log (mg/dL)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
log (mg/dL) | -0.09 [-0.4 to 4.7] | -0.01 [-0.14 to 0.11]

17. Other Pre Specified Outcome: Mean Change in Hemoglobin Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of hemoglobin. The mean changes between baseline, 6 weeks and 12 weeks in hemoglobin with 95% CI were calculated using linear mixed effects model.
Time Frame: baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
g/dL | -0.25 [-0.46 to -0.04] | -0.13 [-0.34 to 0.07]

18. Other Pre Specified Outcome: Mean Change in Plasma Nitrate Over 12 Weeks
Description: A blood sample was drawn for each participant to measure the levels of plasma nitrate. The mean changes between baseline, 6 weeks and 12 weeks in plasma nitrate with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
umol/L | 15.4 [5.9 to 25.0] | -6.3 [-15.7 to 3.1]

19. Other Pre Specified Outcome: Mean Change in Urinary Albumin-to-creatinine Ratios Over 12 Weeks
Description: A urine sample was taken for each participant to measure the levels of urinary albumin-to-creatinine ratios. The mean changes between baseline, 6 weeks and 12 weeks in urinary albumin-to-creatinine ratios with 95% CI were calculated using linear mixed effects model, and the log transformed urinary albumin-to-creatinine ratios was calculated.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: log (mg/g)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
log (mg/g) | 0.04 [-0.27 to 0.36] | 0.02 [-0.29 to 0.33]

20. Other Pre Specified Outcome: Mean Change in Blood Pressure Over 12 Weeks
Description: Blood pressure was measured using the OMRON HEM-907 XL BP Monitor per standard protocol by trained and certified research staff. The mean changes between baseline, 6 weeks and 12 weeks in blood pressure with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
mm Hg
  Systolic blood pressure, mmHg | -2.2 [-6.8 to 2.4] | -0.7 [-5.3 to 3.8]
  Diastolic blood pressure, mmHg | -2.5 [-5.0 to -0.1] | 0.1 [-2.3 to 2.6]

21. Other Pre Specified Outcome: Mean Change in Pulse Over 12 Weeks
Description: Pulse was measured at the brachial artery per standard protocol by trained and certified research staff. The mean changes between baseline, 6 weeks and 12 weeks in pulse with 95% CI were calculated using linear mixed effects model.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Mean Changes Over 12 Weeks (95% CI)
Measure: Mean (95% Confidence Interval); unit: beat/minute
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 35 | 35
beat/minute | 0.6 [-1.7 to 2.3] | -0.5 [-2.8 to 1.9]

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events in the duration of 3 months.
Arm/Group | Treatment | Placebos
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/35
Other Adverse Events (participants affected / at risk) | 11/35 | 14/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=35) | Placebos (N=35)
Serious Adverse Event - Inpatient hospitalization (Cardiac disorders) | 1 (1) | 1 (1) — One SAE in the treatment group included a hospitalization for new onset atrial fibrillation due to a massively dilated left atrium.
OTHER ADVERSE EVENTS (reported when occurring in more than 1.75% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=35) | Placebos (N=35)
Adverse Events (Cardiac disorders) | 11 (55) | 14 (63)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT02552888/Prot_SAP_000.pdf